CLINICAL TRIAL: NCT01796080
Title: The Effect of Simulated Obstructive Apnoea and Hypopnoea on Heart Rhythm in Patients With Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: PAF_V1.1 (05.07.2012)
Record Dates: First submitted 2013-02-18; First posted 2013-02-21 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Patients With Paroxysmal Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mueller manoeuvre (Active Comparator): Mueller manoeuvre lasting for 20 seconds
  Interventions: Other: Mueller manoeuvre
- Inspiratory threshold (Active Comparator): One continuous inspiration through an inspiratory threshold load for 20 seconds
  Interventions: Other: Inspiratory threshold
- Expiratory apnoea (Active Comparator): Expiratory apnoea (without respiratory effort) lasting for 20 seconds
  Interventions: Other: Expiratory apnoea
- Steady state normal breathing (Sham Comparator): Steady state normal breathing for 20 seconds
  Interventions: Other: Steady state normal breathing

INTERVENTIONS:
Other: Mueller manoeuvre
  Arms: Mueller manoeuvre
Other: Inspiratory threshold
  Arms: Inspiratory threshold
Other: Expiratory apnoea
  Arms: Expiratory apnoea
Other: Steady state normal breathing
  Arms: Steady state normal breathing

SUMMARY:
In this randomised controlled cross-over study we will investigate whether intrathoracic pressure changes induced by simulated obstructive apnoea and hypopnoea trigger premature supraventricular and ventricular contractions as well as atrial fibrillation in patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion criteria:

* Age 18-75 years
* History of ECG-documented paroxysmal atrial fibrillation within the last 12 months and currently in sinus rhythm
* Informed consent

Exclusion criteria:

* Mental or physical disability precluding informed consent or compliance with the protocol
* Amiodarone or Dronedarone medication
* Previous radiofrequency ablation for atrial fibrillation
* Severe structural heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with premature myocardial contractions and/or atrial fibrillation | 20 seconds

SECONDARY OUTCOMES:
ECG-derived myocardial de- and repolarization times | 20 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof MD, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Canton of Zurich, Switzerland